CLINICAL TRIAL: NCT05121064
Title: Common Elements Treatment Approach HIV Alcohol Reduction Trial in Zambia
Acronym: CHARTZ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Columbia University (Other); Centre for Infectious Disease Research in Zambia (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Johns Hopkins Bloomberg School of Public Health (Other); University of Zambia (Other)
Responsible Party: Principal Investigator, Michael Vinikoor, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-300008297; P01AA029540 (NIH)
Record Dates: First submitted 2021-11-12; First posted 2021-11-16 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: HIV/AIDS; Alcohol-Related Disorders; Mental Illness
Keywords: HIV; Unhealthy Alcohol Use; Mental Illness; HIV care continuum; sub-Saharan Africa; Alcohol biomarkers; Implementation science
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcohol-Related Disorders; Mental Disorders | interventions — Ethanol; Standard of Care

STUDY DESIGN:
Intervention Model Description: People meeting criteria will be assigned at random to one of 3 study arms.
Who Masked: Investigator
Masking Description: The data manager overseeing data collection and the biostatistician analyzing study outcomes will not be aware of participant study arm until the data are locked for analysis of the primary outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A- Alcohol Brief Intervention (Experimental): Following enrollment and randomization, participants will receive a single session of alcohol brief intervention (BI). Further, standard of care antiretroviral therapy (ART) adherence counseling will be provided as per local guidelines.
  Interventions: Behavioral: Alcohol Brief Intervention
- Arm B- Alcohol Brief Intervention plus Common Elements Treatment Approach (Experimental): Following enrollment and randomization, participants will receive a single session of alcohol brief intervention (BI) and then will be referred to receive Common Elements Treatment Approach (CETA). Further, standard of care antiretroviral therapy (ART) adherence counseling will be provided as per local guidelines. For CETA, a specially trained counselor will contact the participant within 2 weeks of enrollment to arrange for CETA sessions, which occur approximately weekly. Participants will receive 6 to 12 sessions of CETA with the number of sessions based on symptoms and response to therapy.
  Interventions: Behavioral: Alcohol Brief Intervention; Behavioral: Common Elements Treatment Approach
- Arm C- Standard of Care (Active Comparator): Following enrollment and randomization, participants will receive ART adherence counseling, which is the standard of care at the clinics.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Alcohol Brief Intervention — The alcohol brief intervention (BI) was based on CETA'S substance use module and was designed for one-on-one delivery. It is comprised of 6 elements (i.e. assessment, understanding impacts, exploring possibilities of change, goal setting, identifying reasons for alcohol use and skill building) including a 2-week alcohol timeline follow back assessment completed by provider. The alcohol brief intervention (BI) will be conducted by a trained counselor.
  Other Names: BI
  Arms: Arm A- Alcohol Brief Intervention; Arm B- Alcohol Brief Intervention plus Common Elements Treatment Approach
Behavioral: Common Elements Treatment Approach — CETA is a multisession cognitive behavioral therapy (CBT)-based model. CETA consists of elements: engagement, safety assessment, psychoeducation, substance use reduction, behavioral activation, cognitive coping, relaxation, exposure and problem solving. During a weekly clinic meeting, newly enrolled participants who are assigned to get CETA will be assigned to a specific counselor. The counsellor, together with their supervisor, will design an individualized treatment plan including type and order of Common Elements Treatment Approach (CETA) for each participant. The counsellor will contact participants by phone or home visit to schedule CETA session. CETA sessions will begin with standardized clinical monitoring form to track progress of treatment and each session will last 45-90 minutes.
  Other Names: CETA
  Arms: Arm B- Alcohol Brief Intervention plus Common Elements Treatment Approach
Behavioral: Standard of Care — Standard of Care (SOC) at HIV clinics in Zambia consist of Antiretroviral Treatment (ART) adherence counselling. All participants will receive Standard of Care (SOC), but for participants in Arm C it will be the only alcohol treatment. The ART adherence counseling includes brief unstructured discussion of substance use and mental health issues with a focus on issues that reduce adherence and retention issues. ART adherence counseling is delivered in a one-on-one format between patient and counsellor and it usually lasts 5-10 minutes.
  Other Names: SOC
  Arms: Arm C- Standard of Care

SUMMARY:
This study, which is part of the Zambia Alabama HIV Alcohol Comorbidities Program funded by NIH-NIAAA, is designed to examine the efficacy of brief and in-depth cognitive behavioral therapy-based interventions to address, unhealthy alcohol use, comorbid mental health symptoms, and HIV treatment outcomes among people living with HIV in Zambia. A 3-arm trial will be conducted with participants randomized to a brief intervention alone, the brief intervention plus referral to Common Elements Treatment Approach (CETA), or standard of care (SOC).

DETAILED DESCRIPTION:
People with HIV are a priority population for alcohol screening and treatment; however, they may be more likely to underreport their alcohol use and may respond less well to alcohol treatments due to untreated comorbidities. Psychological treatments for unhealthy alcohol use should ideally include components to address common mental health and other substance use comorbidities. However, few current treatments can treat both substance use and mental illness with a single protocol. Further, whether integrated treatment of unhealthy alcohol use and its comorbidities is more effective than alcohol-focused treatment alone needs to be established. There are psychological alcohol treatments that are consider brief interventions (BI), which are time limited and require fewer resources to implement. There are also more complex interventions that require multiple sessions with a provider and are more time and resource intensive; however, they may have more potential for short- and long-term effectiveness.

In this study we will examine the efficacy of both a brief intervention (BI) alone and a more comprehensive and involving the BI followed by Common Elements Treatment Approach (CETA; www.cetaglobal.org) among adults with unhealthy alcohol use and HIV in urban Zambia. CETA is a transdiagnostic cognitive behavioral therapy-based intervention that can flexibly treat a range of conditions including substance use, depression, posttraumatic stress, and anxiety. Further, CETA can be delivered by professional and lay providers. There is already evidence that CETA can reduce alcohol use in the general population in Zambia. In pilot study, the BI plus CETA reduced alcohol use and mental health symptoms more at 6 months than the BI alone. Whether the BI is superior to standard of care (SOC), antiretroviral therapy adherence counseling, is not known.

This study will build on existing knowledge by looking at longer-term effects (12 months) of the interventions, assess impact on HIV outcomes (adherence to antiretrovirals, retention in HIV care, viral suppression), and to understand whether the BI is superior to current SOC. In the study, we will also evaluate implementation factors related to delivery of the two interventions within public sector HIV clinics. Understanding how to implement interventions for unhealthy alcohol use and mental illness is a major priority in the field.

We will have several groups of participants:

* 1 Adults with HIV and unhealthy alcohol use- this group will be enrolled and randomly assigned to one of three Arms (A, B or C) of the study. Arm A will receive alcohol brief intervention (BI), Arm B alcohol brief intervention (BI) plus referral to Common Elements Treatment Approach (CETA), or Arm C standard of care (SOC). The participants in Arm A will receive the single session alcohol brief intervention (BI). Participants in Arm B will also receive the BI and then be referred for CETA, which includes 6-12 sessions with a provider. The participants in Arm C will receive standard of care (SOC) only. All participants will be re-assessed at 6 and 12 months post-enrollment. Patients who participate will provide data on alcohol use, mental health and other substance use comorbidities, and HIV outcomes. Data will be generated through surveys and in some cases through laboratory tests (blood and urine). CETA will be provided by HIV peer counselors, a cadre of lay health worker that supports HIV care delivery at facilities in Zambia.
* 2 CETA counselors- this group will be enrolled and their competency to provide the intervention will be assessed through role plays. Further, they will be included in focus group discussions to understand experiences delivering CETA at HIV clinics.
* 3 Clinic staff- these individuals will be HIV care providers at the study clinics and they will be invited to focus group discussions so we can understand their perspectives on integration of interventions into their clinics.
* 4 Key informants- these are high-level policymakers and HIV and mental health/substance use policy makers and experts in Zambia who can guide us on understanding how to scale up study interventions should they be effective.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Living with HIV
* Receiving HIV care at study site
* Hazardous alcohol use plus at least one mental health or other substance use comorbidity or moderate to severe alcohol use disorder regardless of comorbidity
* 6 months since initiation of Antiretroviral Treatment (ART)
* Suboptimal HIV care outcome based on at least 1 of the following occurences in the past year: Late (at least 14 days from scheduled) Antiretroviral Treatment (ART) drug pick up, HIV viral load (VL) above the limit of assay detection, or referral to enhanced adherence

Exclusion Criteria:

* Plan to relocate out of Lusaka in next 6 months
* No access to a telephone
* Actively suicidal or alcohol intoxication and in need of immediate care
* Currently psychotic
* Participating in another interventional study that would interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 680 (Actual)
Dates: Start 2023-01-24 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
HIV Viral Load Suppression at 6 months | 6 months
  The study will focus on HIV viral load suppression with the definition being HIV RNA concentration below the sensitivity of the assay. In Zambia, it is possible that assays with slightly different HIV RNA sensitivity (for example 20, 40, and 60 copies per milliliter) may be used. Our definition for VLS will be having HIV RNA below the level of the least sensitive assay used during the study. We will estimate and compare risk differences with 95% CIs across the three study arms (i.e. 1=HIV VS and 0=no HIV VS). HIV viral suppression (VS) is the ultimate goal of ART and has individual and public health benefits.

SECONDARY OUTCOMES:
Change in Alcohol Use from enrollment to 6 months | 6 months
  Alcohol use in the study will be measured by the Alcohol Use Disorders Identification Test (AUDIT). The minimum score on the Alcohol Use Disorders Identification Test (AUDIT) is 0 and maximum score on AUDIT is 40. For men, a score of 9 or greater indicates hazardous alcohol consumption. For women a score of 4 or greater indicates hazardous alcohol consumption. Higher AUDIT scores indicate unhealthy alcohol use.
Change in Alcohol Use from enrollment to 12 months | 12 months
  Alcohol use in the study will be measured by the Alcohol Use Disorders Identification Test (AUDIT). The minimum score on the Alcohol Use Disorders Identification Test (AUDIT) is 0 and maximum score on AUDIT is 40. For men, a score of 9 or greater indicates hazardous alcohol consumption. For women a score of 4 or greater indicates hazardous alcohol consumption. Higher AUDIT scores indicate unhealthy alcohol use.
Change in Alcohol Biomarker from enrollment to 6 months | 6 months
  The participant's blood level of phosphatidylethanol (PEth) will be analyzed in several ways. First describe the proportion with alcohol abstinence (PEth <8 ng/ml). Proportion with alcohol abstinence (PEth) level less than 20ng/ml indicate abstinence or light drinking. Second to describe proportion with unhealthy use (PEth>50 ng/ml). Proportion with alcohol abstinence (PEth) level of 20-200ng/ml indicate moderate level of drinking. Higher level of (PEth) indicate hazardous alcohol consumption. Ethl Glucuronide (EtG) will be analyzed to identify to identify patients with false reports of abstinence for exclusion from model.
Change in Alcohol Biomarker from enrollment to 12 months | 12 months
  The participant's blood level of phosphatidylethanol (PEth) will be analyzed in several ways. First describe the proportion with alcohol abstinence (PEth <8 ng/ml). Proportion with alcohol abstinence (PEth) level less than 20ng/ml indicate abstinence or light drinking. Second to describe proportion with unhealthy use (PEth>50 ng/ml). Proportion with alcohol abstinence (PEth) level of 20-200ng/ml indicate moderate level of drinking. Higher level of (PEth) indicate hazardous alcohol consumption. Ethl Glucuronide (EtG) will be analyzed to identify to identify patients with false reports of abstinence for exclusion from model.
Antiretroviral Treatment (ART) Medication Adherence from baseline to 6 months | 6 months
  Antiretroviral Treatment (ART) medication adherence will be assess based on the medication possession ratio (MPR). The medication possession ratio (MPR) metric used characterize engagement in HIV care and is a strong predictor of HIV viral suppression. These data include the date of each medication dispensation and the next scheduled drug pick-up date (based on the number of pills dispensed). MPR will be calculated from ART dispensation data that are extracted at enrollment, 6, and 12 months.
Antiretroviral Treatment (ART) Medication Adherence from enrollment to 12 months | 12 months
  Antiretroviral Treatment (ART) medication adherence will be assess based on the medication possession ratio (MPR). The medication possession ratio (MPR) metric used characterize engagement in HIV care and is a strong predictor of HIV viral suppression. These data include the date of each medication dispensation and the next scheduled drug pick-up date (based on the number of pills dispensed). MPR will be calculated from ART dispensation data that are extracted at enrollment, 6, and 12 months.
Change in HIV Viral Load from enrollment to 6 months | 6 months
  Defined as viral load <1,000 copies at 6 months. Testing will be done by a central lab and results will be returned to the clinic for entry into the patient's medical record so they can be used for clinical care.
Change in HIV Viral Load from enrollment to 12 months | 12 months
  Defined as viral load <1,000 copies at 12 months. Testing will be done by a central lab and results will be returned to the clinic for entry into the patient's medical record so they can be used for clinical care.
Retention in care change from enrollment to 6 months | 6 months
  Defined as being >28 days late for medication at 6 months calculated and compared across trial arms.
Retention in care change from enrollment to 12 months | 12 months
  Defined as being >28 days late for medication at 6 months calculated and compared across trial arms.
Changes in Mental Health and Substance Use from enrollment to 6 months | 6 months
  Changes in mental health, from enrollment to 6 months, based on the PHQ-9 for depression, HTQ for trauma, and GAD-7 for anxiety and changes in non-alcohol substance use based on ASSIST tool and a rapid point-of-care drug test
Changes in Mental Health and Substance Use from enrollment to 12 months | 12 months
  Changes in mental health, from enrollment to 12 months, based on the PHQ-9 for depression, HTQ for trauma, and GAD-7 for anxiety and changes in non-alcohol substance use based on ASSIST tool and a rapid point-of-care drug test
Change in Health Related Quality of Life (QoL) from enrollment to 6 months | 6 months
  Change in health-related Quality of Life (QoL) based on EQ-5D at enrollment and 6 months
Change in Health Related Quality of Life (QoL) from enrollment to 12 months | 12 months
  Change in health-related Quality of Life (QoL) based on EQ-5D at enrollment and 12 months

OTHER OUTCOMES:
Analysis of CETA completion | 12 months
  Common Elements Treatment Approach (CETA) uptake and completion will be tracked. Assessing predictors of treatment completion by estimating a logit model with a binary outcome (1=completer; 0=non-completer). Predictors will be demographic (e.g., sex, age) and clinical factors (e.g., symptom severity).
Process evaluation | 12 months
  A mixed-methods process evaluation with multiple stakeholders will be used to understand how contextual factors impact treatment completion. Quantitative indicators of good implementation are initiation and completion of the brief intervention and CETA, short time from enrollment to first CETA, between CETA sessions, and from enrollment to completion of CETA. High acceptability based on client and provider surveys will also provide quantitative data on the process. In qualitative interviews and focus groups we will discuss quantitative data and gain participant, organizational, and policy perspectives on the results and barriers to optimal implementation.
Cost effectiveness analysis | 12 months
  We will estimate the cost-effectiveness of the Brief Intervention (BI) alone and Brief Intervention + Common Elements Treatment Approach (BI+CETA) compared to Standard of Care (SOC) following standard guidelines. We will calculate incremental cost effectiveness ratios (ICER) comparing each intervention versus its comparator.

CONTACTS AND LOCATIONS:
Locations (3):
- Zambia (3):
  - Chilenje Level 1 Hospital, Lusaka
  - Kalingalinga Health Centre, Lusaka
  - Kamwala Health Centre, Lusaka

REFERENCES:
- [Background] Vinikoor MJ, Sharma A, Murray LK, Figge CJ, Bosomprah S, Chitambi C, Paul R, Kanguya T, Sivile S, Nghiem V, Cropsey K, Kane JC. Alcohol-focused and transdiagnostic treatments for unhealthy alcohol use among adults with HIV in Zambia: A 3-arm randomized controlled trial. Contemp Clin Trials. 2023 Apr;127:107116. doi: 10.1016/j.cct.2023.107116. Epub 2023 Feb 13. PMID 36791907
- [Background] Vinikoor MJ, Sikazwe I, Sharma A, Kanguya T, Chipungu J, Murray LK, Chander G, Cropsey K, Bosomprah S, Mulenga LB, Paul R, Kane J. Intersection of alcohol use, HIV infection, and the HIV care continuum in Zambia: nationally representative survey. AIDS Care. 2023 Oct;35(10):1555-1562. doi: 10.1080/09540121.2022.2092589. Epub 2022 Jun 27. PMID 35761776
- [Background] Figge CJ, Kane JC, Skavenski S, Haroz E, Mwenge M, Mulemba S, Aldridge LR, Vinikoor MJ, Sharma A, Inoue S, Paul R, Simenda F, Metz K, Bolton C, Kemp C, Bosomprah S, Sikazwe I, Murray LK. Comparative effectiveness of in-person vs. remote delivery of the Common Elements Treatment Approach for addressing mental and behavioral health problems among adolescents and young adults in Zambia: protocol of a three-arm randomized controlled trial. Trials. 2022 May 19;23(1):417. doi: 10.1186/s13063-022-06319-4. PMID 35590348
- [Background] Kane JC, Glass N, Bolton PA, Mayeya J, Paul R, Mwenge M, Murray LK. Two-year treatment effects of the common elements treatment approach (CETA) for reducing intimate partner violence and unhealthy alcohol use in Zambia. Glob Ment Health (Camb). 2021 Feb 19;8:e4. doi: 10.1017/gmh.2021.2. eCollection 2021. PMID 34026235
- [Background] Murray LK, Dorsey S, Haroz E, Lee C, Alsiary MM, Haydary A, Weiss WM, Bolton P. A Common Elements Treatment Approach for Adult Mental Health Problems in Low- and Middle-Income Countries. Cogn Behav Pract. 2014 May;21(2):111-123. doi: 10.1016/j.cbpra.2013.06.005. PMID 25620867